CLINICAL TRIAL: NCT05399966
Title: Investigating the Effects of Monarda Didyma Extract Supplementation on Biological Aging of Susceptible Population: a Randomized, Placebo Controlled, Double Blind Parallel Study
Brief Title: Effects of Monarda Didyma Extract Supplementation on Biological Ageing
Acronym: EMODISU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofia Pavanello (Other)
Collaborators: Mibelle AG (Industry)
Responsible Party: Sponsor-Investigator, Sofia Pavanello, Full professor, University of Padova
Organization: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BIOAGELAB202201
Record Dates: First submitted 2022-05-17; First posted 2022-06-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Pilot study; randomized, placebo-controlled, double-blind, parallel design, monocentric.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monarda Didyma extract (Experimental): Monarda Didyma extract
  Interventions: Dietary Supplement: Monarda Didyma extract
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Monarda Didyma extract — Monarda Didyma extract; 100 mg/d. 1capsules/day; daily (1 capsule with the lunch) and plenty of water.
  Arms: Monarda Didyma extract
Dietary Supplement: Placebo — Maltodextrin; 100 mg/d. 1capsules/day; daily (1 capsule with the lunch) and plenty of water.
  Arms: Placebo

SUMMARY:
This research aims to explore the potential benefits of supplementation of a natural ingredient, the Monarda didyma extract, to reduce / delay the biological aging of a susceptible population, thus contributing to two relevant topics in science with important social and economic implications: anti-aging strategies for wellness and healthy aging and environmental sustainability using natural products.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to follow the study protocol procedures to sign the Informed Consent Form prior to screening evaluations
* Age: 45 - 65

Exclusion Criteria:

* Relevant history or presence of any medical disorder potentially interfering with this study (heavy depression, diabetes, active cancer, severe liver disease, heavy cardiovascular disease (e.g., stroke, heart attack))
* Chronic intake of medication/dietary supplements with impact on stress levels (psychologically and physiological)
* Consumption of any dietary/nutritional supplements or functional foods
* Smokers
* High caffeine intake > 5 coffee cups / day
* Gastrointestinal diseases/conditions (ulcerative colitis, Crohn's disease, peptic ulcers, celiac disease)
* Drug-, alcohol- and medication abuses
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Known allergies against the mint family (labiate), especially lemon balm (la cedrella, la melissa, la citronella)
* Pregnancy, breastfeeding or intention to become pregnant during the study
* Participation in another clinical study within the last 4 weeks and concurrent participation in another clinical study
* Blood donation within 4 weeks prior to study start (screening) or during the study
* Anticipating any planned changes in lifestyle for the duration of the study
* Subjects considered inappropriate for the study by investigators, including subjects who are unable or unwilling to show compliance with the protocol

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
DNA methylation age (DNAmAge) | 12 weeks
  DNA methylation age (years)
Age acceleration (AgeAcc) | 12 weeks
  Age acceleration as difference between DNA methylation age and chronological age (years)
Leukocyte telomere length (LTL) | 12 weeks
  Leukocyte telomere length as ratio (T/S) of number telomere repeat sequences (T) to single-copy gene (S)
Mitochondrial DNA copy number (mtDNAcn) | 12 weeks
  Mitochondrial DNA copy number (mtDNAcn) as ratio (MT/S) of mitochondrial DNA copy number (MT) and the singular copy number of a gene (S)

SECONDARY OUTCOMES:
Telomerase expression (∆∆Ct) | 12 weeks
  Telomerase expression as comparative cycle threshold method (∆∆Ct), which compares the difference in cycle threshold values between groups.
Blood pressure | 12 weeks
  Blood pressure as systolic blood and diastolic blood pressure (mm Hg)
Salivary cortisol | 12 weeks
  Salivary cortisol (nmol/L).
Leukocytes | 12 weeks
  Leukocytes (10^9/L)
erythrocytes | 12 weeks
  erythrocytes (10^12/L)
hemoglobin | 12 weeks
  hemoglobin (g/L)
hematocrit | 12 weeks
  hematocrit (L/L)
MCV mean corpuscular volume | 12 weeks
  MCV (fL)
MCH mean corpuscular hemoglobin | 12 weeks
  MCH (pg)
MCHC mean corpuscular hemoglobin concentration | 12 weeks
  MCHC (g/L)
platelets | 12 weeks
  platelets (10^9/L)
C reactive protein | 12 weeks
  C reactive protein - CRP (mg/L)
interleukin 6 | 12 weeks
  interleukin 6 - IL6 (ng/L)
Questionnaire about Quality of Life: World Health Organization's Quality of Life Assessment BREF version (WHOQOL-BREF) | 12 weeks
  Domain scores for the WHOQOL-BREF are calculated by taking the mean of all items included in each domain and multiplying by a factor of four. These scores are then transformed to a 0-100 scale, where 100 is the highest and 0 is the lowest QoL.
Questionnaire about sleeping patterns: Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  The PSQI contains 19 self-reported combined to form seven "component" scores, each of which has a range of 0 (no difficulty) to 3 (severe difficulty) points. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Tracking of Hearth Rate using Miband 6 watch | 12 weeks
  hearth rate as beats per minute (BPM)
Tracking of sleep using Miband 6 watch | 12 weeks
  sleep (hours)
Tracking of mobility using Miband 6 watch | 12 weeks
  mobility (step counts)
Total cholesterol | 12 weeks
  Total cholesterol (mg/dl)
LDL | 12 weeks
  LDL (mg/dl)
HDL | 12 weeks
  HDL (mg/dl)
Triglycerides | 12 weeks
  Triglycerides (mg/dl)
Glycemia | 12 weeks
  Glycemia (mg/dl)
Insulin | 12 weeks
  Insulin (mcU/ml)
HOMA | 12 weeks
  HOMA index - homeostasis model assessment
AST | 12 weeks
  AST (IU/l) aspartate aminotransferase
SGPT | 12 weeks
  SGPT (IU/l) Serum Glutamic Pyruvic Transaminase
GGT | 12 weeks
  GGT (U/l) gamma glutamyl transferase
Creatinine | 12 weeks
  Creatinine (mg/dl)
Waist | 12 weeks
  Waist circumference (cm)
Weight | 12 weeks
  Weight (kg)
Total cholesterol/HDL | 12 weeks
  Total cholesterol/HDL
LDL/HDL | 12 weeks
  LDL/HDL cholesterol ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale Università Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao Q, Lin MT, Zhu YD, Xu HL, Zhao YZ. Recent Trends in Potential Therapeutic Applications of the Dietary Flavonoid Didymin. Molecules. 2018 Oct 6;23(10):2547. doi: 10.3390/molecules23102547. PMID 30301216
- [Background] Feng Z, Pang L, Chen S, Pang X, Huang Y, Qiao Q, Wang Y, Vonglorkham S, Huang Q, Lin X, Wei J. Didymin ameliorates dexamethasone-induced non-alcoholic fatty liver disease by inhibiting TLR4/NF-kappaB and PI3K/Akt pathways in C57BL/6J mice. Int Immunopharmacol. 2020 Nov;88:107003. doi: 10.1016/j.intimp.2020.107003. Epub 2020 Sep 23. PMID 33182043
- [Background] Lin X, Bai F, Nie J, Lu S, Lu C, Zhu X, Wei J, Lu Z, Huang Q. Didymin Alleviates Hepatic Fibrosis Through Inhibiting ERK and PI3K/Akt Pathways via Regulation of Raf Kinase Inhibitor Protein. Cell Physiol Biochem. 2016;40(6):1422-1432. doi: 10.1159/000453194. Epub 2016 Dec 20. PMID 27997902
- [Background] Pavanello S, Campisi M, Tona F, Lin CD, Iliceto S. Exploring Epigenetic Age in Response to Intensive Relaxing Training: A Pilot Study to Slow Down Biological Age. Int J Environ Res Public Health. 2019 Aug 23;16(17):3074. doi: 10.3390/ijerph16173074. PMID 31450859
- [Background] Campisi M, Liviero F, Maestrelli P, Guarnieri G, Pavanello S. DNA Methylation-Based Age Prediction and Telomere Length Reveal an Accelerated Aging in Induced Sputum Cells Compared to Blood Leukocytes: A Pilot Study in COPD Patients. Front Med (Lausanne). 2021 Jul 23;8:690312. doi: 10.3389/fmed.2021.690312. eCollection 2021. PMID 34368190
- [Background] Pavanello S, Campisi M, Fabozzo A, Cibin G, Tarzia V, Toscano G, Gerosa G. The biological age of the heart is consistently younger than chronological age. Sci Rep. 2020 Jul 1;10(1):10752. doi: 10.1038/s41598-020-67622-1. PMID 32612244
- [Background] Pavanello S, Dioni L, Hoxha M, Fedeli U, Mielzynska-Svach D, Baccarelli AA. Mitochondrial DNA copy number and exposure to polycyclic aromatic hydrocarbons. Cancer Epidemiol Biomarkers Prev. 2013 Oct;22(10):1722-9. doi: 10.1158/1055-9965.EPI-13-0118. Epub 2013 Jul 24. PMID 23885040